CLINICAL TRIAL: NCT02251288
Title: A Phase I Randomized Study in Healthy Adults to Assess the Safety, Reactogenicity and Immunogenicity of Priming With an Inactivated A/H7N9 Influenza Virus Vaccine With or Without MF59 Adjuvant Followed by Live Attenuated A/H7N9 Influenza Virus Vaccine
Brief Title: A Phase I Study Priming With an Inactivated A/H7N9 Influenza Virus Vaccine With or Without MF59 Adjuvant Followed by Live Attenuated A/H7N9 Influenza Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 13-0087
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2018-07-01

CONDITIONS: Avian Influenza; Immunisation
Keywords: H7N9 pandemic; inactivated influenza vaccine (pIIV); live attenuated influenza vaccine (pLAIV); MF59 adjuvant
MeSH Terms: conditions — Influenza in Birds | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): 12 patients receive Intramuscular (IM) A/H7N9 15 mcg on Day 1, 12 patients receive A/H7N9 15 mcg plus MF59 adjuvant IM on Day 1 and all receive single dose of Intranasal (IN) sprayer 10^7 FFU H7 N9 pLAIV on Day 29
  Interventions: Biological: Influenza Virus Vaccine, Live Attenuated H7N9 Anhui 2013/AA ca; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Drug: MF59 adjuvant
- Group 2 (Experimental): 12 patients receive A/H7N9 15 mcg IM on Day 1, 12 patients receive A/H7N9 15 mcg plus MF59 adjuvant IM on Day 1 and all receive single dose of IN sprayer10^7 FFU H7 N9 pLAIV on Day 85
  Interventions: Biological: Influenza Virus Vaccine, Live Attenuated H7N9 Anhui 2013/AA ca; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Drug: MF59 adjuvant
- Group 3 (Experimental): 12 patients receive S A/H7N9 15 mcg IM on Day 1, 12 patients receive A/H7N9 15 mcg plus MF59 adjuvant IM on Day 1 and all receive single dose of IN sprayer 10^7 FFU H7 N9 pLAIV on Day 169
  Interventions: Biological: Influenza Virus Vaccine, Live Attenuated H7N9 Anhui 2013/AA ca; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Drug: MF59 adjuvant
- Group 4 (Experimental): 8 patients receive A/H7N9 15 mcg IM on Day 1, 8 patients receive A/H7N9 15 mcg plus MF59 adjuvant IM on Day 1
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Drug: MF59 adjuvant
- Group 5 (Experimental): 12 patients receive A/H7N9 15 mcg plus MF59 adjuvant on Day 1 and Day 29
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Drug: MF59 adjuvant

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Live Attenuated H7N9 Anhui 2013/AA ca — MedImmune supplies pLAIV vaccines as a colorless to pale yellow and clear to slightly cloudy suspension in single, unit-dose, Becton-Dickinson Accuspray™ Nasal Spray Systems sprayer devices. Each filled sprayer device contains a 0.5 mL dose of 10^7FFU of H7N9 Anhui 2013/AA ca vaccine. Group I receives the IN dose on Day 29, Group 2 on Day 85, and Group 3 on Day 169.
  Arms: Group 1; Group 2; Group 3
Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013 — Sanofi supplies the monovalent influenza A/H7N9 virus vaccine as a sterile, clear, and slightly opalescent suspension in single-dose vials containing 15 mcg HA per 0.5 mL. Group 1 through Group5 will receive the IM vaccine on Day 1
Drug: MF59 adjuvant — Novartis supplies the MF59 adjuvant as an oil-in-water milky emulsion in single-use vials containing a fill volume of 0.7 mL. Group 1 through Group 5 will receive MF59 IM on Day 1.

SUMMARY:
A phase I prospective, randomized study in healthy adult subjects at a single center. Adult subjects age 18 to 47 years and meeting all enrollment criteria will choose to participate as subjects who receive inactivated vaccine followed by a live vaccine boost at 4 weeks (Group 1), 12 weeks (Group 2), or 24 weeks (Group 3), or to be in an observational group (Group 4) which will not be scheduled for a booster dose but may serve as a roll-over group for subjects who withdraw prior to the second vaccination but agree to remain in follow-up. A fifth group will receive two intramuscular doses of adjuvanted H7N9 pIIV separated by four weeks. The primary objectives of this study are to (1) assess the safety of H7N9 pLAIV administered to individuals who have previously received MF59-adjuvanted or unadjuvanted H7N9 pIIV, (2) evaluate the ability of a single dose of unadjuvanted H7N9 pIIV to prime for enhanced immunogenicity (booster response) to subsequent administration of antigenically-matched H7N9 pLAIV vaccine, and to (3) evaluate the ability of a single dose of MF59-adjuvanted H7N9 pIIV to prime for enhanced immunogenicity (booster response) to subsequent administration of antigenically-matched H7N9 pLAIV vaccine.

DETAILED DESCRIPTION:
The study will be conducted as a Phase I prospective, randomized study in healthy adult subjects at a single center. Adult subjects age 18 to 47 years and meeting all enrollment criteria will choose to participate as subjects who receive unadjuvanted or adjuvanted H7H9 pIIV vaccine followed by a live vaccine boost at 4 weeks (Group 1, n=24), 12 weeks (Group 2, n=24), or 24 weeks (Group 3, n=24), or to be in an observational group (Group 4, n=16) which will not be scheduled for a booster dose but may serve as a roll-over group for subjects who withdraw prior to the second vaccination but agree to remain in follow-up. Within each group, subjects will be randomized at a 1:1 ratio to receive a single dose of either unadjuvanted H7N9 pIIV at 15 mcg (Subgroup A), or the same vaccine adjuvanted with the oil-in-water emulsion, MF59, (Subgroup B) delivered intramuscularly. Finally, a fifth group (Group 5, n=12) will receive two intramuscular doses of adjuvanted H7N9 pIIV separated by four weeks. The total duration of study participation for all subjects will be approximately 13 months. Recruitment, enrollment and administration of study product will be suspended when one of the following occurs in the clinical or research laboratory at the clinical site: at least two respiratory cultures or PCR assays are determined to be positive for influenza or at least 10% diagnostic tests (rapid tests, respiratory cultures or PCR assays) performed for influenza as positive during two consecutive weeks in the clinical or research laboratory at the clinical site. Recruitment, enrollment and administration of study product may be resumed after 2 weeks without a signal that influenza is still circulating in the community, as defined by the same measures that indicate the start of influenza season (i.e., less than 2 respiratory cultures or PCR assays are determined to positive for influenza or less than 10% of diagnostic tests performed or influenza with positive results). The primary objectives of this study are to (1) assess the safety of H7N9 pLAIV administered to individuals who have previously received MF59-adjuvanted or unadjuvanted H7N9 pIIV, (2) evaluate the ability of a single dose of unadjuvanted H7N9 pIIV to prime for enhanced immunogenicity (booster response) to subsequent administration of antigenically-matched H7N9 pLAIV vaccine, and to (3) evaluate the ability of a single dose of MF59-adjuvanted H7N9 pIIV to prime for enhanced immunogenicity (booster response) to subsequent administration of antigenically-matched H7N9 pLAIV vaccine. The secondary objectives of this study are to (1) assess the safety of priming with MF59-adjuvanted H7N9 pIIV or unadjuvanted H7N9 pIIV, (2) assess the immune response in subjects vaccinated with a single dose of MF59-adjuvanted H7N9 pIIV or a single dose of unadjuvanted H7N9 pIIV, and to (3) compare the booster effect seen after intervals of 4 weeks, 12 weeks, or 24 weeks within each priming group.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures, including future use of specimens.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant, non-breastfeeding females, 18 to 47 years old, inclusive.
4. Are in good health, as determined by medical history, and targeted physical examination to ensure any existing medical diagnoses or conditions (except those exclusionary) are stable* **.

   *Stable chronic medical condition - no change in prescription medication, dose, or frequency of medication in the last 3 months (defined as 90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months (defined as 180 days). Any change that is due to change of health care provider, insurance company etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion.

   **Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Note: Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subject Exclusion Criteria), vitamins, and contraceptives are permitted.
5. Oral temperature is less than 100.4 degrees Fahrenheit.
6. Pulse is 55 to 100 bpm, inclusive.
7. Systolic blood pressure is 90 to 140 mmHg, inclusive.
8. Diastolic blood pressure is 55 to 90 mmHg, inclusive.
9. Women of childbearing potential* in sexual relationships with men must use an acceptable method of contraception** from 30 days prior to pIIV administration until 90 days after last study vaccination.

   *Not sterilized via tubal ligation, bilateral oophorectomy or hysterectomy and still menstruating or < 1 year of the last menses if menopausal).

   **Includes, but is not limited to, abstinence from intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, and licensed hormonal methods, with use of a highly effective method of contraception for a minimum of 30 days prior to study product exposure and agree to practice highly effective contraception for the duration of study product exposure, including 3 months (defined as 90 days) after the last study vaccination. A highly effective method of contraception is defined as one which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
10. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness within 72 hours prior to study vaccination.
2. Any medical disease or condition that, in the opinion of the investigator, is a contraindication to study participation*.

   *Includes medical disease or condition that would place the subject at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or their successful completion of the study.
3. Have history of any significant acute or chronic medical conditions* or need for chronic medications that, in the opinion of the investigator, will interfere with immunogenicity or affect safety.

   *Chronic medical condition - a medical condition persisting 3 months (defined as 90 days) or longer
4. Have immunosuppression or are taking systemic immunosuppressants as a result of an underlying illness or treatment.
5. Diagnosis of asthma or reactive airway disease within the past 2 years.
6. History of surgical splenectomy.
7. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 36 months prior to vaccination.
8. Have known active neoplastic disease or a history of any hematologic malignancy.
9. Have known hepatitis B or hepatitis C infection.
10. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
11. Known allergy or intolerance to oseltamivir.
12. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
13. Have a history of Guillain-Barré Syndrome.
14. Have a history of neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to study vaccination.
15. Have a history of autoimmune disease*.

    *Including, but not limited to, neuroinflammatory diseases, vasculitis, clotting disorders, dermatitis, arthritis, thyroiditis, or muscle, liver, or kidney disease.
16. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
17. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
18. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
19. Have taken oral or parenteral corticosteroids of any dose within 30 days prior to study vaccination.
20. Chronic use (defined as daily use for > 7days within the 30 days prior to study vaccination) of any inhaled medication, including inhaled corticosteroids.
21. Received any licensed live vaccine within 30 days prior to pIIV vaccination. This is inclusive of licensed seasonal influenza vaccines.
22. Received any licensed inactivated vaccine within 14 days prior to pIIV vaccination. This is inclusive of licensed seasonal influenza vaccines.
23. Planned receipt of any vaccine from the first study vaccination through the follow-up visit at approximately 56 days after the second study vaccination. This is inclusive of licensed seasonal influenza vaccines
24. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
25. Received an experimental agent* within 30 days prior to pIIV administration or planned receipt of an experimental agent to within 90 days after pLAIV administration.

    *Includes vaccine, drug, biologic, device, blood product, or medication.
26. Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period.

    *Includes trials that have a study intervention such as a drug, biologic, or device
27. Prior participation in a clinical trial of influenza A/H7 vaccine* or have a history of A/H7 actual or potential exposure or infection prior to the first study vaccination.

    *Documented receipt of placebo in such a trial is not exclusionary
28. Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) in the time between the first study vaccination and 56 days after the second study vaccination.
29. Positive screening pregnancy test or other evidence of pregnancy.
30. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after their last study vaccination.
31. Seropositive to the H7N9 influenza A virus (serum HAI titer > 1:8) during the screening period prior to the first study vaccination.
32. Positive urine drug screen for opiates and cocaine at the time of check-in for the period of confinement.
33. Positive ELISA and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1) during the screening period prior to vaccination.
34. Current smoker unwilling to stop smoking for the period of confinement. A nicotine patch during the period of confinement may be offered.

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers determined by neuraminidase inhibiting antibody by enzyme-linked lectin assay (ELLA) | Day 29
Geometric mean titers determined by neuraminidase inhibiting antibody by enzyme-linked lectin assay (ELLA) for Group 2 | Day 113
Geometric mean titers determined by neuraminidase inhibiting antibody by enzyme-linked lectin assay (ELLA) for Group 3 | Day 197
Geometric mean titers determined by neuraminidase inhibiting antibody by enzyme-linked lectin assay (ELLA) for Groups 1, 5 | Day 57
Occurrence of respiratory reactogenicity following pLAIV vaccination for Group 1 | Day 29 through Day 39
Occurrence of respiratory reactogenicity following pLAIV vaccination for Group 2 | Day 85 through Day 95
Occurrence of respiratory reactogenicity following pLAIV vaccination for Group 3 | Day 169 through Day 179
Occurrence of solicited systemic reactogenicity following pLAIV vaccination for Group 1 | Day 29 through Day 39
Occurrence of solicited systemic reactogenicity following pLAIV vaccination for Group 2 | Day 85 through Day 95
Occurrence of solicited systemic reactogenicity following pLAIV vaccination for Group 3 | Day 169 through Day 179
Occurrence of study vaccine-related serious adverse events following pLAIV vaccination for Group 1 | Day 29 through Day 209
Occurrence of study vaccine-related serious adverse events following pLAIV vaccination for Group 2 | Day 85 through Day 265
Occurrence of study vaccine-related serious adverse events following pLAIV vaccination for Group 3 | Day 169 through Day 349
Occurrence of study vaccine-related unsolicited non-serious adverse events following pLAIV vaccination for Group 1 | Day 29 through Day 57
Occurrence of study vaccine-related unsolicited non-serious adverse events following pLAIV vaccination for Group 2 | Day 85 through 113
Occurrence of study vaccine-related unsolicited non-serious adverse events following pLAIV vaccination for Group 3 | Day 169 through 197
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 2 | Day 113
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 3 | Day 197
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Groups 1, 5 | Day 57
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) for Group 2 | Day 113
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) for Group 3 | Day 197
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) for Groups 1,5 | Day 57
Percentage of subjects shedding vaccine virus as detected by rRT-PCR following pLAIV vaccination for Group 1 | Day 29 through Day 36
Percentage of subjects shedding vaccine virus as detected by rRT-PCR following pLAIV vaccination for Group 2 | Day 85 through Day 92
Percentage of subjects shedding vaccine virus as detected by rRT-PCR following pLAIV vaccination for Group 3 | Day 169 through Day 176
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells | Day 29
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 2 | Day 113
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 2 | Day 141
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 2 | Day 265
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 3 | Day 197
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 3 | Day 225
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Group 3 | Day 349
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Groups 1, 5 | Day 209
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Groups 1, 5 | Day 57
Percentage of subjects with positive B cell responses by plasmablast assays on peripheral blood mononuclear cells for Groups 1, 5 | Day 85

SECONDARY OUTCOMES:
Geometric mean titers of serum HAI antibody | Day 1
Geometric mean titers of serum HAI antibody | Day 29
Geometric mean titers of serum HAI antibody for Group 2 | Day 113
Geometric mean titers of serum HAI antibody for Group 2 | Day 141
Geometric mean titers of serum HAI antibody for Group 2 | Day 265
Geometric mean titers of serum HAI antibody for Group 3 | Day 197
Geometric mean titers of serum HAI antibody for Group 3 | Day 225
Geometric mean titers of serum HAI antibody for Group 3 | Day 349
Geometric mean titers of serum HAI antibody for Groups 1, 5 | Day 209
Geometric mean titers of serum HAI antibody for Groups 1, 5 | Day 57
Geometric mean titers of serum HAI antibody for Groups 1, 5 | Day 85
Geometric mean titers of serum NtAb antibody | Day 1
Geometric mean titers of serum NtAb antibody | Day 29
Geometric mean titers of serum NtAb antibody for Group 2 | Day 113
Geometric mean titers of serum NtAb antibody for Group 2 | Day 141
Geometric mean titers of serum NtAb antibody for Group 2 | Day 265
Geometric mean titers of serum NtAb antibody for Group 3 | Day 197
Geometric mean titers of serum NtAb antibody for Group 3 | Day 225
Geometric mean titers of serum NtAb antibody for Group 3 | Day 349
Geometric mean titers of serum NtAb antibody for Groups 1, 5 | Day 209
Geometric mean titers of serum NtAb antibody for Groups 1, 5 | Day 57
Geometric mean titers of serum NtAb antibody for Groups 1, 5 | Day 85
Occurrence of adverse events of special interest following pIIV vaccination | Day 1 through Day 366
Occurrence of adverse events of special interest following pIIV vaccination for Group 5 | Day 1 through Day 394
Occurrence of local reactogenicity following pIIV vaccination | Day 1 through Day 8
Occurrence of local reactogenicity following pIIV vaccination for Group 5 | Day 29 through Day 36
Occurrence of new-onset chronic medical conditions for Group 2 | Day 1 through Day 265
Occurrence of new-onset chronic medical conditions for Group 3 | Day 1 through Day 349
Occurrence of new-onset chronic medical conditions for Group 4 | Day 1 through Day 181
Occurrence of new-onset chronic medical conditions for Groups 1, 5 | Day 1 through Day 209
Occurrence of study vaccine-related serious adverse events following pIIV vaccination | Day 1 through Day 366
Occurrence of study vaccine-related serious adverse events following pIIV vaccination for Group 5 | Day 29 through Day 394
Occurrence of study vaccine-related unsolicited non-serious adverse events following pIIV vaccination | Day 29
Occurrence of study vaccine-related unsolicited non-serious adverse events following pIIV vaccination for Group 5 | Day 57
Occurrence of systemic reactogenicity following pIIV vaccination | Day 1 through Day 8
Occurrence of systemic reactogenicity following pIIV vaccination for Group 5 | Day 29 through Day 36
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine | Day 1
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine | Day 29
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 1, 5 | Day 209
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 1, 5 | Day 85
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 2 | Day 141
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 2 | Day 265
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 3 | Day 225
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H7N9 antigen contained in the study vaccine for Group 3 | Day 349
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines | Day 1
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines | Day 29
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 2 | Day 113
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 2 | Day 141
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 2 | Day 265
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 3 | Day 197
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 3 | Day 225
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Group 3 | Day 349
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Groups 1, 5 | Day 209
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Groups 1, 5 | Day 57
Percentage of subjects achieving a serum NtAb titer of 1:40 or greater against the H7N9 antigen contained in the study vaccines for Groups 1, 5 | Day 85
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) | Day 29
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Group 2 | Day 141
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Group 2 | Day 265
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Group 3 | Day 225
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Group 3 | Day 349
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Groups 1, 5 | Day 209
Percentage of subjects achieving seroconversion (a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer = / > 1:40 or a pre-vaccination HAI titer = / > 1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer) for Groups 1, 5 | Day 85
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) | Day 29
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 2 | Day 113
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 2 | Day 141
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 2 | Day 265
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 3 | Day 197
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 3 | Day 225
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Group 3 | Day 349
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Groups 1, 5 | Day 209
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Groups 1, 5 | Day 57
Percentage of subjects achieving seroconversion (a pre-vaccination NtAb titer <1:10 and a post-vaccination NtAb titer = / > 1:40 or a pre-vaccination NtAb titer = / > 1:10 and a minimum 4-fold rise in post-vaccination NtAb titer) for Groups 1, 5 | Day 85

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York, United States